CLINICAL TRIAL: NCT06004830
Title: Feasibility, Acceptability, and Preliminary Efficacy of Off-Label Medications for Alcohol Use Disorder Among Patients With HIV: An Open-Label Pilot Study
Brief Title: Off-Label Medications for Alcohol Use Disorder Among Patients With HIV: Pilot Study 1
Acronym: HARP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000033919_a; 1P01AA029545-01 (NIH)
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Use Disorder; Hiv
MeSH Terms: conditions — Alcoholism; Acquired Immunodeficiency Syndrome | interventions — Spironolactone

STUDY DESIGN:
Intervention Model Description: Single arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Spironolactone (Experimental): Participants will receive a prescription for spironolactone
  Interventions: Drug: Spironolactone

INTERVENTIONS:
Drug: Spironolactone — All participants will receive a prescription for spironolactone and will meet with a clinical pharmacist and addiction psychiatrist for further support

SUMMARY:
This study seeks to determine the feasibility, acceptability, and preliminary efficacy of an intervention consisting of off-label use of a medication with strong efficacy data for alcohol use disorder (AUD) with medical management and a clinical pharmacist-delivered behavioral intervention in reducing alcohol use among individuals with HIV and AUD.

DETAILED DESCRIPTION:
This is a series of three open-label pilot studies that consist of a 12-week intervention including off-label use of medication with MM and a clinical pharmacist-delivered behavioral intervention to treat AUD. Participants will receive counseling that incorporates brief feedback and advice with motivational enhancement techniques to assist the participant in changing their behaviors with respect to alcohol consumption and/or polypharmacy defined as taking five or more medications, particularly if those medications interact with alcohol. In addition, participants will be offered spironolactone in the first pilot study. The rationale for utilizing an open-label pilot study design is to determine the feasibility, acceptability, safety, and preliminary efficacy of this intervention for the management of AUD. Participants will be interviewed with regards to their perspectives on feasibility and acceptability. They will be instructed to have medication bottles at study visits to assess medication adherence and will be assessed with readiness to change metrics and questions regarding quantity and frequency of alcohol use. Patients will also be asked to complete an AUDIT-C screen and the Alcohol Symptom Checklist at the start of the study period to screen for mild, moderate, or severe AUD. Several assessments including interviews and laboratory testing will be done at study visits.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with HIV
* Receive care at the Atlanta VA Healthcare System
* Age 18 or over
* Meet criteria for mild, moderate, or severe alcohol use disorder by the DSM-5 Alcohol Symptom Checklist and the Alcohol Use Disorders Identification Test-Consumption (AUDIT-C) screen
* Have evidence of significant alcohol use: PEth > 20ng/ml
* Prescribed >=5 medications
* Have cell phone or reliable contact number
* Can provide written informed consent

Exclusion Criteria:

* Active engagement in formal alcohol treatment including medications for alcohol use disorder at the time of enrollment
* Self-report or laboratory test confirming pregnancy, nursing, or trying to conceive
* Life-threatening or unstable medical, surgical, or psychiatric condition that prohibits participation (including current or past intent to harm oneself or others within the prior 12 months and not receiving treatment
* Untreated moderate to severe opioid use disorder
* Residence out of state
* Inability to read or understand English
* History of serious hypersensitivity or adverse reaction to study medication
* Taking potentially interactive medication(s): eplerenone, potassium supplementation, lithium, digoxin, cholestyramine, heparin and low-molecular weight heparin for spironolactone)
* Hyperkalemia defined as serum potassium ≥ 5.0 mEq/L on the most recent laboratory test performed in the past 60 days prior to enrollment or Addison's disease or estimated glomerular filtration rate <50 mL/min/1.73 m2 (for spironolactone)
* Creatinine level of ≥1.5 mg/dl (for spironolactone)
* Already prescribed the pilot medication at the time of study recruitment.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who complete enrollment and duration of sessions | 12 weeks
  Proportion of participants who complete enrollment and duration of sessions to assess feasibility of study
Number of sessions completed | 12 weeks
  Number of sessions completed to assess acceptability of study
Adherence to Medication | 12 weeks
  Medication adherence will be measured by the number of prescriptions filled by electronic health record to assess acceptability of study
Safety of study assessed by adverse events reporting | 12 weeks
  Safety will be assessed by the percentage of study participants who report adverse events

SECONDARY OUTCOMES:
Efficacy of study - change in self-reported alcohol use | 12 weeks
  Change in self-reported alcohol use (# of days of alcohol use and # of drinks per day) on the Timeline Followback.
Efficacy of study - change in PEth (phosphatidylethanol) results | 12 weeks
  PEth is a biomarker for alcohol consumption. Change in PEth result from baseline PEth levels.

CONTACTS AND LOCATIONS:
Overall Officials: E. Jennifer Edelman, MD, MHS, Principal Investigator — Yale University
Locations (1):
- Atlanta VA Medical Center, Decatur, Georgia, United States